CLINICAL TRIAL: NCT00903344
Title: Impact of Vitamin D Supplementation on Lactation Associated Bone Loss
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Leigh Eck, MD (Other)
Collaborators: Bio-Tech Pharmacal, Inc. (Industry)
Responsible Party: Sponsor-Investigator, Leigh Eck, MD, Assistant Professor, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 11711
Record Dates: First submitted 2009-05-14; First posted 2009-05-18 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2014-08-18 (Estimated); Status verified 2014-08

CONDITIONS: Osteoporosis
MeSH Terms: conditions — Osteoporosis | interventions — Cholecalciferol; Geritol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D (Experimental): 4000IU Vitamin D3 in tablet taken daily with multivitamin
  Interventions: Drug: Vitamin D3
- Multivitamin (Active Comparator): Multivitamin with 400IU vitamin D tablet
  Interventions: Dietary Supplement: Multivitamin

INTERVENTIONS:
Drug: Vitamin D3 — 4000IU vitamin D3 tablet taken daily
  Arms: Vitamin D
Dietary Supplement: Multivitamin — Multivitamin containing 400IU vitamin D in tablet taken daily
  Arms: Multivitamin

SUMMARY:
Studies have shown that lactation is associated with a loss of bone density from four to seven percent at the spine and hip among women who lactate for six months. Decline in bone density with lactation occurs rapidly. Although bone density increases after weaning, there is controversy on whether or not it is completely restored. Epidemiological studies find no significant negative impact of lactation on bone mass or fractures, and in fact there is evidence that lactation has a positive effect on bone mass. We think that interventions that attenuate this physiologic loss of bone that is associated with lactation and accelerate restoration of bone mass after weaning may result in improved long term bone mass and diminished fracture risk.

DETAILED DESCRIPTION:
Adequate vitamin D stores are necessary for skeletal health. Vitamin D deficiency is pronounced in women of child bearing age as well as pregnant women in the United States. This study will provide important information about whether vitamin D supplementation may positively impact the normal physiologic loss of bone mass that is observed during lactation.

Recruitment will begin while subjects are pregnant in order to expedite entry into the study in the immediate post-partum period. If subjects are deemed eligible during pregnancy, contact information to include name, address, expected delivery date and two contact phone numbers will be obtained. Subjects will be contacted two weeks prior to expected delivery date and then again at expected delivery date. Subjects will be followed for a total of 18 months.

ELIGIBILITY:
Inclusion Criteria:

* Fully lactating mothers age 18 and up
* Within 1 month after delivery
* Plan to breast feed for at least 6 months

Exclusion Criteria:

* Known metabolic bone disease
* Chronic renal insufficiency
* Chronic corticosteroid use
* Eating disorder
* Estrogen containing hormonal contraception use
* Daily use of >400IU Vitamin D supplementation
* Delivery of Multiples
* Delivery of a singleton with a birth weight of <2500 grams
* Preterm delivery of baby
* History of kidney stones

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2009-12; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leigh Eck, MD, Principal Investigator — University of Kansas Medical Center
Locations (1):
- University of Kansas Medical Center, Kansas City, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Vitamin D - Experimental: 4000IU Vitamin D3 in tablet taken daily with multivitamin
  Vitamin D3: 4000IU vitamin D3 tablet taken daily
- Multivitamin - Active Comparator: Multivitamin with 400IU vitamin D tablet
  Multivitamin: Multivitamin containing 400IU vitamin D in tablet taken daily
Period: Overall Study
Arm/Group | Vitamin D - Experimental | Multivitamin - Active Comparator
Started | 12 | 10
3 Month Visit | 10 | 10
6 Month Visit | 9 | 10
Completed | 7 | 7
Not Completed | 5 | 3
Not completed — Pregnancy | 2 | 3
Not completed — Lost to Follow-up | 3 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Vitamin D - Experimental | Multivitamin - Active Comparator | Total
Number analyzed (Participants) | 12 | 10 | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 29 (6) | 32 (3) | 30 (4.64)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 10 | 22
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 10 | 22

OUTCOME MEASURES:

1. Primary Outcome: Change in Bone Mineral Density (BMD) in HIP at 6 Months
Time Frame: Change from Baseline to 6 months
Measure: Mean (Standard Deviation); unit: grams/cm^2
Arm/Group | Vitamin D - Experimental | Multivitamin - Active Comparator
Number analyzed (Participants) | 9 | 10
grams/cm^2 | -0.041 (0.014) | 0.011 (0.122)

2. Secondary Outcome: Change in 25-hyroxyvitamin D Levels at 3 Months
Description: Difference in means between visits
Time Frame: Change from Baseline to 3 Months
Population: At 3 month visit there had been two participants that dropped out in the Vitamin D - Experimental group. No participants had dropped out in the Multivitamin - Active Comparator group but the test for this specific outcome measure for two of the groups' participants was not included in the results.
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Vitamin D - Experimental | Multivitamin - Active Comparator
Number analyzed (Participants) | 10 | 8
ng/ml | 2.600 (7.230) | -5.850 (7.713)

3. Secondary Outcome: Change in 25-hyroxyvitamin D Levels at 6 Months
Time Frame: Change from Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: ng/ml
Arm/Group | Vitamin D - Experimental | Multivitamin - Active Comparator
Number analyzed (Participants) | 9 | 10
ng/ml | 1.889 (7.865) | -3.200 (13.774)

4. Secondary Outcome: Change in Bone Mineral Density (BMD) at HIP at 3 Months
Time Frame: Change from Baseline to 3 months
Population: At 3 month visit there had been two participants that dropped out in the Vitamin D - Experimental group. No participants had dropped out in the Multivitamin - Active Comparator group but the test for this specific outcome measure for one of the group's participants was not included in the results.
Measure: Mean (Standard Deviation); unit: grams/cm^2
Arm/Group | Vitamin D - Experimental | Multivitamin - Active Comparator
Number analyzed (Participants) | 10 | 9
grams/cm^2 | -0.017 (0.009) | -0.016 (0.022)

5. Secondary Outcome: Change in Bone Mineral Denisty (BMD) in SPINE at 3 Months
Description: difference in mean
Time Frame: Change from Baseline to 3 Months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: grams/cm^2
Arm/Group | Vitamin D - Experimental | Multivitamin - Active Comparator
Number analyzed (Participants) | 10 | 9
grams/cm^2 | -0.025 (0.071) | -0.025 (0.030)

6. Secondary Outcome: Change in Bone Mineral Denisty (BMD) in SPINE at 6 Months
Description: difference in the mean
Time Frame: Change from Baseline to 6 Months
Measure: Mean (Standard Deviation); unit: grams/cm^2
Arm/Group | Vitamin D - Experimental | Multivitamin - Active Comparator
Number analyzed (Participants) | 9 | 10
grams/cm^2 | -0.060 (0.036) | -0.109 (0.115)

ADVERSE EVENTS:
Arm/Group | Vitamin D - Experimental | Multivitamin - Active Comparator
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/10
Other Adverse Events (participants affected / at risk) | 1/12 | 0/10
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Vitamin D - Experimental (N=12) | Multivitamin - Active Comparator (N=10)
Constipation (Gastrointestinal disorders) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes